CLINICAL TRIAL: NCT05520437
Title: Omega-3 Fatty Acids Supplementation on Stress-induced Changes to Kynurenine Metabolism and Mood in Physically Active and Inactive Males
Brief Title: Effect of Omega-3 Fatty Acids on Kynurenine Metabolism and Mood
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Medical University of Gdansk (Other)
Collaborators: National Science Centre, Poland (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2019/35/N/NZ7/03757
Record Dates: First submitted 2021-07-14; First posted 2022-08-30 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: Stress-induced Mood; Kynurenine Pathway and Its Metabolites
Keywords: Omega-3; Kynurenine pathway
MeSH Terms: interventions — Fatty Acids, Omega-3

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physically active males (Experimental): Half of the study population will consist of long-distance runners with 2-5 years of experience in running and similar times in covering the half-marathon distance.
  Interventions: Dietary Supplement: Omega-3 fatty acids; Dietary Supplement: Placebo
- Physically inactive males (Experimental): The other half of the study population will consist of age-matched individuals involved in no regular physical activity.
  Interventions: Dietary Supplement: Omega-3 fatty acids; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Omega-3 fatty acids — Participants received Omega-3 supplements (NAMEDSPORT) in the form of softgels over a period of 12 weeks. The supplement is certified by the International Fish Oil Standards™ (IFOS™) Program. Daily dose contained a total of 3276 mg of Omega 3 (4000 mg of fish oil of which: EPA 2234mg; DHA 916mg).
Dietary Supplement: Placebo — Participants will receive a placebo in the form of MCT oil capsules with no effect on the hypothesized outcome.

SUMMARY:
The purpose of the current study is to explore the effect of omega-3 fatty acids supplementation on stress-induced changes to kynurenine metabolism and mood.

The objectives of this research project are as follows:

1. To compare biochemical parameters (KYN and KYNA, markers of oxidative stress, and markers of inflammation) between physically active and inactive males
2. To determine the impact of a 3-month supplementation with omega-3 fatty acids on mood, inflammation markers and oxidative stress, and changes in KYN and KYNA
3. To determine the impact of the stress manipulation test (TSST) on mood and changes in KYN and KYNA before and after the omega-3 fatty acids supplementation

DETAILED DESCRIPTION:
The purpose of the current study is to explore the effect of omega-3 fatty acids supplementation on stress-induced changes to kynurenine metabolism and mood. While previous studies suggest that peripheral tryptophan conversion to KYN is activated by stress and inflammatory factors, the evidence is based on animal models only. Hence, this will be the first study to test this phenomenon on humans. Omega-3 fatty acids supplementation in this study aims to reduce the inflammatory factors. The stress response in participants will be experimentally controlled by conducting a stress manipulation task. Finally, based on the findings that exercise-induced PGC-1α expression in skeletal muscles might protect against stress-induced neurobiological mechanisms of depressed mood, the study will compare two groups of participants: passive individuals and physically active individuals who might have higher activity of KAT in skeletal muscles. This study design will allow to investigate the effect of long-term endurance training on L-kynurenine levels and mood. Considering a constant rise in the consumed ratio of omega-6/omega-3 as well as a more sedentary lifestyle and higher experienced stress in western countries, this study could have a great therapeutic potential and will expand our understanding of mechanisms of how diet and exercise can influence mood.

The objectives of this research project are as follows:

1. To compare biochemical parameters (KYN, KYNA, markers of oxidative stress, and inflammation) between physically active and inactive males
2. To determine the impact of a 3-month supplementation with omega-3 fatty acids on changes in the kynurenine and kynurenic acid
3. To determine the impact of a 3-month supplementation with omega-3 fatty acids on inflammation markers and oxidative stress
4. To determine the impact of a 3-month supplementation with omega-3 fatty acids on mood
5. To determine the impact of the stress manipulation test (TSST) on kynurenine metabolism before and after the omega-3 fatty acids supplementation

Procedure

Prior to the study, participants will be outlined the study protocol and will be assured about the right to withdrawn at any time. Following this, a written informed consent will be obtained from all participants.

Before the start of the intervention blood samples will be collected from the participants to determine the percentage content of omega-3 fatty acids in the serum and red blood cell, KYN and KYNA, markers of oxidative stress (lipid peroxidation products, protein carbonyls), and inflammation markers (CRP, IL-10, TNF). Mood will be assessed using validated psychological measures: Mood Adjective Check List (UMACL) and the Depression, Anxiety and Stress Scale - 21 Items (DASS-21). This will be followed by inducing a stress response with a validated stress manipulation test, the Trier Social Stress Test (TSST) in both groups of participants. After the stress manipulation test, mood and biological parameters will be reassessed.

All participants will receive omega-3 supplementation for the period of 12 weeks.

12 weeks after the start of the intervention blood samples will be collected from the participants to determine the omega-3 fatty acid levels, KYN and KYNA, markers of oxidative stress (lipid peroxidation products, protein carbonyls), and inflammation markers (CRP, IL-10, TNF). Mood will be assessed using UMACL and DASS. This will be followed by inducing a stress response (TSST) in both groups of participants. Straight after the stress manipulation test, and 1 hour after the stress manipulation test, mood and biological parameters will be reassessed.

ELIGIBILITY:
Inclusion Criteria:

* long-distance runners with 2-5 years of experience in running and similar times in covering the half-marathon distance
* age-matched individuals involved in no regular physical activity
* must provide a signed informed consent form

Exclusion Criteria:

* DSM-5 psychiatric diagnoses other than depression and anxiety disorders (American Psychiatric Association, 2013)
* neurological disorders any other serious medical problems
* taking dietary supplements

Ages: 28 Years to 48 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-11-20 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Kynurenine pathway and its metabolites | 3 months
  Before the intervention and 12 weeks after the start of the intervention blood samples will be collected from the participants to determine kynurenine pathway and its metabolites, namely Xanthurenic acid [ng/mL], Kynurenic acid [ng/mL], Kynurenine [ng/mL] and 3-Hydroxykynurenine [ng/mL]. This will be followed by inducing a stress response with the Trier Social Stress Test (TSST) in both groups of participants. Straight after TSST and one hour after the stress manipulation test Xanthurenic acid [ng/mL], Kynurenic acid [ng/mL], Kynurenine [ng/mL] and 3-Hydroxykynurenine [ng/mL] will be reassessed.

SECONDARY OUTCOMES:
Mood | 3 months
  Mood Adjective Check List (UMACL) will be used to assess mood (Mathews, Chamberlain & Jones, 1990, adapted to Polish by Ewa Goryńska, 2005). UMACL measures mood in three dimensions of the core affect: Tense Arousal (minimum value: 9, maximum value: 36), Energetic Arousal (minimum value: 10, maximum value: 40), and Hedonic Tone (minimum value: 10, maximum value: 40), with higher scores representing higher levels of the mood dimensions.
Mood | 3 months
  The Depression, Anxiety and Stress Scale - 21 Items (DASS-21) will be used to assess mood. DASS-21 measures the emotional states of depression, anxiety and stress (for each of the subscales the minimum value is 10 and the maximum value is 42, with higher scores representing higher levels of the emotional states).
Omega-3 fatty acids | 3 months
  The percentage content of omega-3 fatty acids in the blood will be assessed (1) before the intervention (2) 12 weeks after the start of the intervention, (3) following the stress manipulation test (Trier Social Stress Test (TSST)), (4) and one hour after TSST.
Inflammation markers | 3 months
  C-reactive protein (CRP) [mg/l] levels will be assessed (1) before the intervention (2) 12 weeks after the start of the intervention, (3) following the stress manipulation test (Trier Social Stress Test (TSST)), (4) and one hour after TSST.
Oxidative stress | 3 months
  Lipid peroxidation products levels will be assessed (1) before the intervention (2) 12 weeks after the start of the intervention, (3) following the stress manipulation test (Trier Social Stress Test (TSST)), (4) and one hour after TSST.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Gdańsk, Gdansk, Poland

REFERENCES:
- [Derived] Bidzan-Wiacek M, Tomczyk M, Blazek M, Mika A, Antosiewicz J. No Effects of Omega-3 Supplementation on Kynurenine Pathway, Inflammation, Depressive Symptoms, and Stress Response in Males: A Placebo-Controlled Trial. Nutrients. 2024 Oct 31;16(21):3744. doi: 10.3390/nu16213744. PMID 39519577
- [Derived] Tomczyk M, Bidzan-Wiacek M, Kortas JA, Kochanowicz M, Jost Z, Fisk HL, Calder PC, Antosiewicz J. Omega-3 fatty acid supplementation affects tryptophan metabolism during a 12-week endurance training in amateur runners: a randomized controlled trial. Sci Rep. 2024 Feb 19;14(1):4102. doi: 10.1038/s41598-024-54112-x. PMID 38374149